CLINICAL TRIAL: NCT04870814
Title: Comparison of 4 Tactical Tourniquets Used in War Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020PPRC05; 2021-A00049-32 (Other: IDRCB)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hemorrhage
Keywords: Tactical tourniquet
MeSH Terms: conditions — Hemorrhage | interventions — Ultrasonography; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: All the participants will test the 4 tourniquets (1 tourniquet model = 1 arm) both as a "fitter" (the person who set up the tourniquet) and as a "receiver" (the person on whom the tourniquet is applied).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SOFTT® Gen 4 tactical tourniquet (Active Comparator): The SOFTT® Gen 4 (Tactical Medical Solutions, Anderson) tactical tourniquet will be assessed.
  Interventions: Device: Tactical tourniquet set up; Diagnostic Test: Medical ultrasound; Other: Questionnaire
- CAT® Gen 7 tactical tourniquet (Active Comparator): The CAT® Gen 7 (C-A-T® Resources, Rock Hill) tactical tourniquet will be assessed.
  Interventions: Device: Tactical tourniquet set up; Diagnostic Test: Medical ultrasound; Other: Questionnaire
- SAM XT® tactical tourniquet (Active Comparator): The SAM XT® (SAM Medical Products®, Wilsonville) tactical tourniquet will be assessed.
  Interventions: Device: Tactical tourniquet set up; Diagnostic Test: Medical ultrasound; Other: Questionnaire
- RMT® 1.5 tactical tourniquet (Active Comparator): The RMT® 1.5 (m2®, Winooski) tactical tourniquet will be assessed.
  Interventions: Device: Tactical tourniquet set up; Diagnostic Test: Medical ultrasound; Other: Questionnaire

INTERVENTIONS:
Device: Tactical tourniquet set up — The tactical tourniquet will be set up to the upper limb and the lower limb during a maximum of 2 minutes.
Diagnostic Test: Medical ultrasound — The efficacy of tactical tourniquet set up will be assessed by medical ultrasound.
Other: Questionnaire — The participants will have to fill a questionnaire assessing pain (for the "receiver"), ease of use, stability and rusticity (for the "fitter").

SUMMARY:
Bleeding remains the leading cause of death in combat, and the literature suggests that tourniquetable hemorrhage is the second leading cause of preventable death, behind non- tourniquetable hemorrhage.

Currently, most Western armed forces recommend the use of the tactical tourniquet in combat for the management of tourniquetable hemorrhage.

The SOFTT® tourniquet (Tactical Medical Solutions, Anderson) is the tactical tourniquet currently in use by the French armed forces. As the contract will soon come to an end, the question of its renewal arises.

The purpose of this study is to compare 4 commercially available tactical tourniquets in healthy volunteers.

The hypothesis of the research is that one of the 4 tourniquets compared is faster to set up than the others.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Student of the Military Health School of Lyon Bron (Ecoles Militaires de Santé de Lyon Bron; EMSLB);
* Periodic medical examination up to date with the mention "fitness for duty";
* Holder of the "Combat Rescue Level 1" training.

Exclusion Criteria:

* Vascular pathology;
* Current progressive pathology of any kind;
* History of thrombo-embolic disease;
* Presence of cardiovascular risk factors (diabetes, hypertension, dyslipidemia, smoking > 1 cigarette/day, BMI > 25);
* Iliofemoral and axillary vascular abnormalities detected by systematic Doppler ultrasound;
* Presence of symptoms suggestive of COVID-19;
* Positive COVID-19 antigen test;
* In contact with a person diagnosed positive for COVID-19 within 15 days prior to inclusion;
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Time required to apply the tactical tourniquet. | Each day during 4 consecutive days
  The tourniquet application time, in seconds, measured with a stopwatch. The stopwatch will be started when the fitter takes the tourniquet, pre-positioned in a tourniquet pouch on his bullet vest.
  The stopwatch will be stopped as soon as at least one of the following conditions is verified
  * the fitter judges the fitting to be effective
  * the fitter cannot tighten any more (technical limit)
  * the tourniquet is too painful for the receiver.

SECONDARY OUTCOMES:
Occlusion of the downstream arterial flow following after tactical tourniquet application | Each day during 4 consecutive days
  The occlusion of the downstream arterial flow will be assessed by medical ultrasound after tactical tourniquet application
Ease of use of the tactical tourniquet | Each day during 4 consecutive days
  The ease of use of the tactical tourniquet will be measured via a 5-point scale: "very easy", "easy", "intermediate", "hard" and "very hard".
Rusticity of the tactical tourniquet | Each day during 4 consecutive days
  The rusticity of the tactical tourniquet will be assessed via a questionnaire: "sufficiently rustic" or "not sufficiently rustic"
Stability of the tactical tourniquet | Each day during 4 consecutive days
  The stability of the tactical tourniquet will be assessed via a questionnaire, on a 5-point scale: "unstable", "not very stable", "moderately stable", "stable" or "extremely stable".
Pain experienced by the receiver during application of the tactical tourniquet | Each day during 4 consecutive days
  Pain experienced by the receiver during application of the tactical tourniquet, measured by a scale ranging from 0 (no pain) to 10 (most unbearable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Desgenettes, Lyon, France